CLINICAL TRIAL: NCT01996020
Title: Intraoperative Trans-fontanel Cerebral Ultrasonography in Infants During Pediatric Cardiac Surgery Under Cardiopulmonary Bypass
Brief Title: Measurement of Cerebral Flow Using Transfontanellar Doppler in Infants Under Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Assistant professor, Seoul National University Hospital
Other Study IDs: H-1208-018-421
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Transfontanellar Doppler can measure the velocity at both the carotid artery and the anterior cerebral artery during cardiopulmonary bypass in congenital heart disease patients. This study can provide reference value of appropriate cerebral blood flow velocity during pediatric cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. the patients less than 1 year of age undergo congenital heart surgery with cardiopulmonary bypass
2. written informed consent is obtained from their guardians in accordance with the requirements of the local ethics committee

Exclusion Criteria:

1. synostosis
2. skull abnormality or fracture
3. epidural hematoma, scalp hematoma

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with congenital heart disease scheduled to recieve cardiac surgery under CPB
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
cerebral blood flow velocity | 6hour
  during cardiac surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park YH, Song IK, Lee JH, Kim HS, Kim CS, Kim JT. Intraoperative trans-fontanellar cerebral ultrasonography in infants during cardiac surgery under cardiopulmonary bypass: an observational study. J Clin Monit Comput. 2017 Feb;31(1):159-165. doi: 10.1007/s10877-015-9815-3. Epub 2015 Dec 21. PMID 26691513